CLINICAL TRIAL: NCT00778414
Title: Randomized, Open - Label, 2 - Way Crossover, Bioequivalence Study of Amoxicillin-Clavulanic Acid 600mg - 42.9 mg/ 5 mL Oral Suspension and Augmentin ES - 600 (Reference) Following a 600 mg - 42.9 mg Dose in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Amoxicillin-Clavulanic Acid 600 mg - 42.9 mg/ 5 mL Oral Suspension Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 60249
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence Amoxicillin Clavulanic acid 600mg 42.9 mg per 5 mL oral suspension
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Amoxicillin-Clavulanic acid 600mg - 42.9 mg/ 5 mL oral suspension of ranbaxy
  Interventions: Drug: Amoxicillin-Clavulanic acid 600mg - 42.9 mg/ 5 mL oral suspension
- 2 (Active Comparator): Augmentin ES - 600
  Interventions: Drug: Amoxicillin-Clavulanic acid 600mg - 42.9 mg/ 5 mL oral suspension

INTERVENTIONS:
Drug: Amoxicillin-Clavulanic acid 600mg - 42.9 mg/ 5 mL oral suspension

SUMMARY:
The objective of this study was to compare the rate and extent of absorption Ranbaxy Laboratories Limited, India, amoxicillin - clavulanic acid and GlaxoSmithKline, U.S.A. (Augmentin ES-600), amoxicillin - clavulanic acid, administered as a 1 x 5 mL (600 mg - 42.9 mg) oral suspension, under fasting conditions.

DETAILED DESCRIPTION:
This was a single center, randomized, single-dose, open-label, 2 - way crossover bioequivalence study to compare the rate and extent of absorption of a test amoxicillin - clavulanic acid versus Augmentin ES - 600, a reference amoxicillin - clavulanic acid, under fasting condition. Prior to study commencement, subjects were randomly assigned to a treatment in accordance with the randomization scheme generated by Anapharm. Subjects were confined to the Anapharm Clinical Research Facility from at least 10 hours prior to the drug administration until after the 12 - hour post dose blood draw, in each period. The treatment phases were separated by a washout period of 20 days.

A total of 55 healthy, adult subjects signed the study - specific Informed Consent Form and were confined for Period I; of these subjects, 48 (24 males and 24 females) were enrolled and were dosed in the study; 42 of these enrolled subjects completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in this study will be members of the community at large. The recruitment advertisements may use various media types (e.g. radio, newspaper, SFBC Anapharm Web site, SFBC Anapharm volunteers' database). Subjects must meet all of the following criteria to be included in the study:

  1. Male or female, smoker or non - smoker, 18 years of age or older
  2. Capable of consent
  3. BMI should be greater than, or equal to 19.0 and less than 30.0

Exclusion Criteria:

* Subjects to whom any of the following applies will be excluded from the study:

  1. Clinically significant illness or surgery within 4 weeks prior to dosing
  2. Any clinically significant abnormality or abnormal laboratory test results found during medical screening
  3. Any reason which, in the opinion of the Clinical Sub - Investigator, would prevent the subjects from participating in the study
  4. Positive test for hepatitis B, hepatitis C or HIV at screening
  5. ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening
  6. History of significant alcohol abuse or drug abuse within one year prior to the screening
  7. Regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [ 1 unit = 150 mL of wine, 360 mL of beer, 0r 45 mL of 40% alcohol])
  8. Use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to the screening visit or positive urine drug screen at screening
  9. History of allergic reactions to amoxicillin - clavulanic acid, penicillin, or other related drugs
  10. Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, Omeprazole; examples of inhibitors: antidepressants (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolines, antihistamines) within 30 days prior to administration of the study medication
  11. Use of an investigational drug or participation in an investigational study within 30 days prior to dosing
  12. Clinically significant history or presence of any gastrointestinal pathology (e.g.: chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g.: diarrhea, vomiting) liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug.
  13. Any clinically significant history or presence of neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, or metabolic disease
  14. Use of the prescription medication within 14 days prior to the administration of study medication or over - the - counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to the administration of the study medication, except for topical products without systemic absorption and hormonal contraceptives
  15. Difficulty to swallow the study medication
  16. Smoking more than 25 cigarettes per days
  17. Any food allergy, intolerance, restriction or special diet that, in the opinion of the Clinical Sub-Investigator, could contraindicate the subject's participation in this study
  18. A depot injection or an implant of any drug (other than hormonal contraceptives) within 3 months prior to administration of the study medications
  19. Donation of plasma (500 mL) within 7 days prior to the drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures for this study) prior to administration of the study medication as follows:
* 50 mL to 599 mL of whole blood within 30 days
* More than 499 ml of whole blood within 56 days prior to the drug administration t) Wear of dentures or presence of braces at the time of dosing or any piercing in mouth, lips, and/ or tongue u) Positive urine pregnancy test at screening v) Breast feeding subject w) Female subjects of child bearing potential having unprotected sexual intercourse with any non - sterile male partner (i.e. male who have not been sterilized by vasectomy for at least 6 months) within 14 days prior to study drug administration. Hormonal contraceptives are permitted during the study but are not an acceptable method of contraception. Acceptable methods of contraception are:
* intra-uterine contraceptive device (placed at least 4 weeks prior to study drug administration)
* Condom or diaphragm + spermicide

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-06; Primary Completion 2006-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Anapharm, Québec, Quebec, Canada

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html